CLINICAL TRIAL: NCT05241808
Title: Girls Can...Move! Testing the Feasibility of a Community-based Physical Activity Intervention for Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deirdre Dlugonski (Other)
Responsible Party: Sponsor-Investigator, Deirdre Dlugonski, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 59680
Record Dates: First submitted 2022-01-05; First posted 2022-02-16 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Physical Inactivity
Keywords: physical literacy; female; accelerometer; exercise
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No-treatment group that only participates in pre- and post-testing.
- Experimental (Experimental): Experimental group participants will receive the 8-week Girls Can...Move! program.
  Interventions: Behavioral: Girls Can...Move!

INTERVENTIONS:
Behavioral: Girls Can...Move! — Girls Can...Move! is an 8-week intervention designed to increase physical literacy and physical activity among middle school aged girls. One-hour, in-person sessions will be held twice per week for a total of 16 sessions. Each session involves: a brief educational lesson related to physical activity participation, a 30-minute group physical activity session, and a take-home challenge. The physical activities will prioritize enjoyment of physical activity and promote the development of movement competence. These activities may include: yoga; Zumba; Pilates; strength training; kick boxing; circuit training; etc.
  Arms: Experimental

SUMMARY:
The purpose of this research is to learn about how to promote physical activity among adolescent girls by testing the feasibility and initial effectiveness of the Girls Can...Move! intervention. Girls Can...Move! will target each component of physical literacy by providing opportunities for adolescent girls to gain knowledge about their own physical activity level, to explore and practice different types of physical activities, and to learn from active female role models. Female participants (n = 30) from one middle school will be randomly assigned to the Girls Can...Move! intervention group or a control group at a 1:1 ratio. The primary outcome variables, physical activity and physical literacy, will be assessed before and after the 8-week Girls Can...Move! intervention using accelerometers and online surveys.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Enrolled in 6th, 7th, or 8th grade at target school

Exclusion Criteria:

* Engage in 60 minutes of moderate-to-vigorous physical activity on more than 3 days per week
* Doctor has told child/parent that there are certain types of activities that the child should not do
* Preexisting injuries or health conditions that limit physical activity

Ages: 11 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Participants must identify as female.
Enrollment: 17 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Girls Can...Move! intervention | pre-intervention (week 0)
  The number of participants enrolled, intervention session attendance (experimental group only), and participant satisfaction with intervention (experimental group only) will be included as feasibility measures.
Change in physical activity | pre-intervention immediately following 8-week intervention period (week 9)
  Participants will wear an Actigraph accelerometer to measure change in physical activity from pre- to post- intervention for the experimental compared to control group.
Change in physical literacy | pre-intervention (week 0) and immediately following 8-week intervention period (week 9)
  Participants will complete measures of self-reported physical literacy (PLAYself survey) at pre- and post-intervention to measure change in perceived physical literacy between experimental and control groups.

SECONDARY OUTCOMES:
Change in peer social support | pre-intervention (week 0) and immediately following 8-week intervention period (week 9)
  Participants will complete measures of self-reported peer social support at pre- and post-intervention to measure change in perceived social support between experimental and control groups.
Change in parental social support | pre-intervention (week 0) and immediately following 8-week intervention period (week 9)
  Participants will complete measures of self-reported parental social support at pre- and post-intervention to measure change in perceived social support between experimental and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No